CLINICAL TRIAL: NCT05431036
Title: Evaluation of a Combined Model of Lung Aeration Score and Diaphragmatic Indices by Transthoracic Ultrasonography in Predicting Weaning Success in Critically Ill Patients.
Brief Title: Evaluation of a Combined Model in Predicting Weaning Outcome in Critically Ill Patients.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Mohammed Taghyan, Assistant lecturer, chest department,Principal Investigator,Clinical Professor, Assiut University
Other Study IDs: lung US in ICU patient
Record Dates: First submitted 2022-06-12; First posted 2022-06-24 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Weaning Failure
Keywords: LUS; DUS; RSBI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: transthoracic ultrasonography — 1. The lung ultrasound score (LUS) will be calculated according to the observed worst ultrasound pattern and Finally, the LUSs of all the parts will added to obtain the total LUS for each patient (maximum36 points)
  2. The diaphragmatic ultrasound will performed for assessment of diaphragmatic thickness and motion.

SUMMARY:
The purpose of our study is to assess lung aeration and diaphragmatic indices by transthoracic ultrasonography in patients ready to be weaned from mechanical ventilation as predictors of weaning success

DETAILED DESCRIPTION:
Assessment of lung aeration and diaphragmatic indices by transthoracic ultrasonography in patients ready to be weaned from mechanical ventilation as predictors of weaning success in critically ill patients .

ELIGIBILITY:
Inclusion Criteria:

* Patients more than18 years old.
* All patients intubated and requiring mechanical ventilation for 48 hours or more at respiratory intensive care unit (RICU)
* Patients fullfiled the criteria of readiness to wean according to European Respiratory Society guidelines (ERS)

Exclusion Criteria

* Patients with neuromuscular disease or diaphragmatic paralysis.
* Patients with tracheostomy.
* Patients who undergone surgical operations especially abdominal and thoracic operation.
* Patients with diseases that may affect the diaphragm (including pneumothorax, pneumomediastinum, patients with inserted intercostal tube (ICT), third trimester of pregnancy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study group will be mechanically ventilated for at least 48 hours. Patients will be assessed daily for fulfillment of criteria of readiness to wean according to European Respiratory Society guidelines and assessment of the three parameters which is Rapid shallow breathing index ( RSBI), lung ultrasound score( LUS) and Diaphragmatic ultrasound (DUS) will be done for predicting weaning success.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of lung aeration by lung ultrasound score using MEDESION SONOACE R3 portable ultrasound apparatus in patients ready to be weaned from mechanical ventilation (MV) as a predictor of weaning success. | baseline
  The lung ultrasound score (LUS) will be calculated according to the observed worst ultrasound pattern using the convex probe (MEDESION SONOACE R3 portable ultrasound, Korea 2010). (normal aeration, LUS = 0);( moderate loss of lung aeration (multiple, well-defined B lines), LUS = 1);( severe loss of lung aeration (multiple coalescent B lines), LUS = 2); (lung consolidation, LUS = 3).Finally, the LUSs of all the parts will added to obtain the total LUS for each patient (maximum36 points).
Assessment of diaphragmatic thickness by diaphragmatic ultrasonography M-mode in patients ready to be weaned from MV as a predictor of weaning success. | baseline
  The diaphragmatic ultrasound will performed for assessment of diaphragmatic thickness by M-Mode Using the high frequency linear probe of 7.5 MHz.This will done in serial manner beginning 24 hours after RICU admission,then during spontaneous breathing trial till the patient is liberated from mechanical ventilation. DT difference (DTD) will be calculated by subtracting The Diaphragm thickening fraction (DTF) will calculated as: DTD/(DT at end-expiration) × 100%
Assessment of diaphragmatic motion by diaphragmatic ultrasonography M-mode in patients ready to be weaned from MV as a predictor of weaning success. | baseline
  The diaphragmatic ultrasound will performed for assessment of diaphragmatic motion by M-mode using the curvilinear low frequency probe (5 MHz).This will done in serial manner beginning 24 hours after RICU admission,then during spontaneous breathing trial till the patient is liberated from mechanical ventilation. Diaphragmatic excursion (DE) will identified and measured. DE amplitude will measured on the vertical axis by tracing from the baseline to the point of maximum height of inspiration on the graph.

SECONDARY OUTCOMES:
Compare between sonographic lung aeration assessment, diaphragmatic indices and rapid shallow breathing index(RSBI) as predictors for results of weaning from mechanical ventilation(MV) | baseline
  Compare between sonographic lung aeration assessment, diaphragmatic indices and RSBI as predictors for results of weaning from MV and showing the predictive value for which parameter to predict weaning sucess alone or combining all three parameters together.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa M Taghyan, Ass.Lecturer, Principal Investigator — Chest department at Assuit university hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Matamis D, Soilemezi E, Tsagourias M, Akoumianaki E, Dimassi S, Boroli F, Richard JC, Brochard L. Sonographic evaluation of the diaphragm in critically ill patients. Technique and clinical applications. Intensive Care Med. 2013 May;39(5):801-10. doi: 10.1007/s00134-013-2823-1. Epub 2013 Jan 24. PMID 23344830
- [Background] Soummer A, Perbet S, Brisson H, Arbelot C, Constantin JM, Lu Q, Rouby JJ; Lung Ultrasound Study Group. Ultrasound assessment of lung aeration loss during a successful weaning trial predicts postextubation distress*. Crit Care Med. 2012 Jul;40(7):2064-72. doi: 10.1097/CCM.0b013e31824e68ae. PMID 22584759
- [Background] Li S, Chen Z, Yan W. Application of bedside ultrasound in predicting the outcome of weaning from mechanical ventilation in elderly patients. BMC Pulm Med. 2021 Jul 9;21(1):217. doi: 10.1186/s12890-021-01605-4. PMID 34243739